CLINICAL TRIAL: NCT06118502
Title: A Clinical Trial of Adaptive Treatment for Early Smoking Cessation Relapse
Acronym: ADAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tracy Smith, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 00128175; 1R01CA284649-01 (NIH)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cigarette Smoking; Smoking Behaviors; Treatment
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Intervention Model Description: An Adaptive, Multi-Randomization Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adaptive Randomization 1 (Experimental): This arm includes people who did not respond to 4 weeks of pharmacotherapy (either varenicline or combination NRT). After a 4-week course of pharmacotherapy, participants that are not responding to medication will receive four weeks of the other FDA approved option, either varenicline or combination NRT, with instructions to try to quit again
  Interventions: Behavioral: Switching to a different medication
- Non-Adaptive Randomization 1 (Experimental): This arm includes people who did not respond to 4 weeks of pharmacotherapy (either varenicline or combination NRT). After a 4-week course of pharmacotherapy, participants that are not responding to the medication will receive four additional weeks of the same medication with instructions to try to quit again
  Interventions: Behavioral: Continued use of the same medication
- Harm Reduction Randomization 2 (Experimental): This arm includes people who did not respond to two 4-week courses of pharmacotherapy (either varenicline or combination NRT or both). After two 4-week courses of pharmacotherapy, participants who are not responding to medication will be randomly assigned to a harm reduction group (e-cigarettes). Participants assigned to the harm reduction group will receive four weeks of e-cigarette product with instructions to switch completely
  Interventions: Behavioral: Switching to a harm reduction tobacco product
- Non-Adaptive Randomization 2 (Experimental): This arm includes people who did not respond to two 4-week courses of pharmacotherapy (either varenicline or combination NRT or both sequentially). After two four-week courses of pharmacotherapy, participants that are not responding to the medication will receive four additional weeks of the same medication with instructions to try to quit again.
  Interventions: Behavioral: Continued use of the same medication

INTERVENTIONS:
Behavioral: Switching to a different medication — Participants will receive four weeks of the other FDA approved option, either varenicline or combination NRT, with instructions to try to quit again at week 4.
  Arms: Adaptive Randomization 1
Behavioral: Continued use of the same medication — Participants will receive four additional weeks of the same medication (varenicline or NRT) with instructions to try to quit again at week 4.
  Arms: Non-Adaptive Randomization 1; Non-Adaptive Randomization 2
Behavioral: Switching to a harm reduction tobacco product — Participants will receive four weeks of e-cigarette products with instructions to switch completely at Week 8
  Arms: Harm Reduction Randomization 2

SUMMARY:
This is a research study to find out if treatment decision making can be improved for smokers who find it difficult to quit with medications. Everyone who participates in this study will receive free product, either nicotine replacement therapies (patches and lozenges), varenicline, or a harm reduction product (e-cigarette) for a full 12 weeks. Most participants will receive some combination of these treatments, depending on individual response to each.

All visits and study assessments will be entirely remote. All treatments will be provided free of charge for the first 12 weeks. After that, the study team will contact the participants 6 months after the first study phone call to complete another survey. The study lasts six months and will involve 8 surveys.

DETAILED DESCRIPTION:
Treatment seeking smokers across both Alabama and South Carolina (N=544) will be recruited and consented through established online methods and randomized to receive a 4-week course of either varenicline or combination NRT (patch + lozenge), counterbalanced. Using a concrete and measurable indicator of early treatment success (3 days non-smoking), smokers demonstrating early success at 4 week follow-up will continue with another four weeks of same medication, either varenicline or combination NRT. Those who do not demonstrate early success will be randomized to a subsequent 4-week course of either a) continuation of same medication, or b) switch to the other FDA approved option, either varenicline or combination NRT. The same process will repeat at Week 8, wherein treatment responders will continue with their ongoing medication and non-responders will be randomized to a final 4-week course of either a) continuation of same medication or b) switch to an e-cigarette. End of treatment outcomes will be assessed at Week 12 at which time no more product will be offered. Final follow-up at Week 24 will ascertain all primary (cessation) and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who want to quit

Exclusion Criteria:

* Non-smokers

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Non-responders after initial course of FDA-approved medication | 8 weeks
  7-day point prevalence abstinence at Week 8 among non-responders at Week 4

SECONDARY OUTCOMES:
Dependence and duration of longest quit attempt | 12 weeks
  7-day point prevalence abstinence at Week 12 among non-responders at Week 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No